CLINICAL TRIAL: NCT04685941
Title: Treatment of Slow-flow After Primary Percutaneous Coronary Intervention With Flow-mediated Hyperemia
Acronym: RAIN FLOW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación EPIC (Other)
Collaborators: Barcicore-Lab (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPIC24-RAIN-FLOW
Record Dates: First submitted 2020-12-22; First posted 2020-12-28 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Coronary Microvascular Disease; Myocardial Infarction
Keywords: Coronary Microvascular Disease; Myocardial Infarction
MeSH Terms: conditions — Microvascular Angina; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug-mediated hyperemia (Other): Patients presenting with slow flow after PPCI undergo to at least 200 mcg of intracoronary nitroprussiate or 500 mcg of intracoronary adenosine during 2 minutes
  Interventions: Drug: Drug-mediated hyperemia
- Flow-mediated hyperemia (Experimental): Patients presenting with slow flow after PPCI undergo to controlled saline intracoronary infusion by a dedicated microcatheter (RayFlow) at 20 ml/min during 2 minutes
  Interventions: Other: Flow-mediated hyperemia

INTERVENTIONS:
Drug: Drug-mediated hyperemia — Intracoronary bolus of at least 200 mcg of nitroprussiate or 500 mcg of intracoronary adenosine during 2 minutes. Operators are allowed to combine both drugs.
  Arms: Drug-mediated hyperemia
Other: Flow-mediated hyperemia — Intracoronary saline infusion at 20 ml/min via dedicated microcatheter (RayFlow; Hexacath, France) during two minutes.
  Arms: Flow-mediated hyperemia

SUMMARY:
A total of 100 patients with ST-elevation myocardial infarction (STEMI) presenting slow-flow after primary-percutaneous coronary intervention (PPCI) will be randomized to pharmacologic treatment with hyperemic drugs versus flow-mediated hyperemia.

DETAILED DESCRIPTION:
Slow-flow phenomena is observed around 15% of patients undergoing PPCI and has been associated with poor prognosis. Hyperemic drugs, such as nitroprussiate and adenosine, have not yet demonstrated to reduce the infarct size and prognosis in patients with slow flow. Controlled flow-mediated hyperemia using a dedicated catheter for intracoronary saline infusion has been shown to stimulate microcirculatory vasodilatation in stable patients similarly as hyperemic drugs.

The aims of the study are to compare the absolute microcirculatory resistance of the infarct-related artery presenting with slow flow after PPCI, as assessed by intracoronary thermo-dilution, treated with standard pharmacologic hyperemia versus flow-mediated hyperemia; and to compare the angiographic TIMI frame count after treatment of slow flow phenomena with the two investigated strategies.

ELIGIBILITY:
Inclusion Criteria:

1. ST elevation myocardial infarction Killip I <12 hours since symptoms onset.
2. ST elevation > 2 mm anterior leads or > 1 mm inferior or lateral leads.
3. Sustained slow coronary flow (TIMI flow 0-2) for at least 30 seconds after stent implantation or stent post-dilatation.

Exclusion Criteria:

1. Previous myocardial infarction in the culprit artery
2. Previous stroke
3. Advanced kidney disease (creatinine clearance <30 ml / min).
4. Active bleeding
5. Allergy to contrast, nitroprussiate or adenosine.
6. Culprit lesion in coronary bypass, left main coronary artery or stent thrombosis
7. Macroscopic thrombus embolization in the infarct-related artery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Angiographic TIMI frame count | 2 minutes
  Cine-fluoroscopic recording of the infarct-related artery (IRA) at 30 frames/second and off-line core-laboratory assessment of the number of cineframes needed for dye to reach standardized distal landmarks is the coprimary endpoint. Long TIMI frame counts are indicative of slow coronary flow. Previous studies showed TIMI frame counts of 30 (SD 12) after nitroprussiate in slow flow STEMI patients. The present study is powered to assess 25 percent difference between study groups (80 percent power and 5 percent alfa error).
Minimal microcirculatory resistance (MMR) | 2 minutes
  MMR is assessed by intracoronary thermodilution with a dedicated pressure wire and microcatheter (RayFlow, Hexacath) during saline infusion at 20 ml/min. MMR is measured offline by the core-laboratory at 20 seconds of the saline infusion in the standard medical treatment group and at 2 minutes and 20 seconds in the experimental group. According to previous studies, MMR was 537 Wood units (SD 289). The present study is powered to assess 30 percent difference between study groups after study intervention (80 percent power and 5 percent alfa error).
Comparison of the MMR in the experimental group during the two-minutes saline infusion | 2 minutes
  Experimental treatment with saline infusion via microcatheter is performed continuously recording the pressure and temperature values of the culprit artery. Off-line core-laboratory assessment of the MMR will be performed at 20 seconds and at 2 minutes of the saline infusion.
Comparison of the Absolute coronary flow between the study groups. | 2 minutes
  Absolute coronary flow is performed simultaneously with the MMR. This value shows the coronary blood flow of the culprit artery during maximal hyperemia.

CONTACTS AND LOCATIONS:
Locations (5):
- Spain (5):
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitario Puerta del Mar, Cadiz
  - Hospital La Princesa, Madrid

REFERENCES:
- [Background] Ndrepepa G, Tiroch K, Keta D, Fusaro M, Seyfarth M, Pache J, Mehilli J, Schomig A, Kastrati A. Predictive factors and impact of no reflow after primary percutaneous coronary intervention in patients with acute myocardial infarction. Circ Cardiovasc Interv. 2010 Feb 1;3(1):27-33. doi: 10.1161/CIRCINTERVENTIONS.109.896225. Epub 2010 Jan 26. PMID 20118156
- [Background] Airoldi F, Briguori C, Cianflone D, Cosgrave J, Stankovic G, Godino C, Carlino M, Chieffo A, Montorfano M, Mussardo M, Michev I, Colombo A, Maseri A. Frequency of slow coronary flow following successful stent implantation and effect of Nitroprusside. Am J Cardiol. 2007 Apr 1;99(7):916-20. doi: 10.1016/j.amjcard.2006.10.057. Epub 2007 Feb 12. PMID 17398183
- [Background] Wijnbergen I, van 't Veer M, Lammers J, Ubachs J, Pijls NH. Absolute coronary blood flow measurement and microvascular resistance in ST-elevation myocardial infarction in the acute and subacute phase. Cardiovasc Revasc Med. 2016 Mar;17(2):81-7. doi: 10.1016/j.carrev.2015.12.013. Epub 2016 Jan 7. PMID 26905054
- [Background] van 't Veer M, Adjedj J, Wijnbergen I, Toth GG, Rutten MC, Barbato E, van Nunen LX, Pijls NH, De Bruyne B. Novel monorail infusion catheter for volumetric coronary blood flow measurement in humans: in vitro validation. EuroIntervention. 2016 Aug 20;12(6):701-7. doi: 10.4244/EIJV12I6A114. PMID 27542781
- [Background] Gibson CM, Schomig A. Coronary and myocardial angiography: angiographic assessment of both epicardial and myocardial perfusion. Circulation. 2004 Jun 29;109(25):3096-105. doi: 10.1161/01.CIR.0000134278.50359.CB. No abstract available. PMID 15226226
- [Derived] Gomez-Lara J, Gracida M, Rivero F, Gutierrez-Barrios A, Muntane-Carol G, Romaguera R, Fuentes L, Marcano A, Roura G, Ferreiro JL, Teruel L, Brugaletta S, Alfonso F, Comin-Colet J, Gomez-Hospital JA. Treatment of Slow-Flow After Primary Percutaneous Coronary Intervention With Flow-Mediated Hyperemia: The Randomized RAIN-FLOW Study. J Am Heart Assoc. 2023 Jul 4;12(13):e030285. doi: 10.1161/JAHA.123.030285. Epub 2023 Jun 22. PMID 37345805